CLINICAL TRIAL: NCT04905680
Title: GluCoach - Technology-enabled Lifestyle Intervention Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Collaborators: Health Promotion Board, Singapore (Other Government)
Responsible Party: Principal Investigator, Dr Falk Mueller-Riemenschneider, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Glucoach
Record Dates: First submitted 2021-05-19; First posted 2021-05-28 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Pre-diabetes
Keywords: Lifestyle coaching; mHealth
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: This is an experimental-control study design where up to 260 individuals at risk of developing diabetes (blood glucose levels of 6.1 to 6.9 mmol/L) will be randomly allocated to the experimental and control groups (1:1 randomization).
  Participants in the control group will not receive any health coaching and are not required to carry out any study activities after they have completed the baseline lifestyle tracking session. At the end of the study, they will attend a 20- to 30-minute session with a coach to have their baseline lifestyle tracking results explained to them and receive personalised suggestions on lifestyle modifications.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The health screening before the study and at the end of study will collect anthropometric data (height, weight, waist and hip circumference), blood pressure data, and blood samples (for testing of HbA1c, fasting blood glucose, fasting insulin and lipid profile). Individuals are provided with an educational brochure upon receiving their screening results. Participants will then go through a baseline lifestyle tracking session using a study-issued smartphone and smartwatch, pre-installed with certain study applications. For participants in the control arm, there is no health coaching or study activities until the end of the study, where individuals will attend a 20- to 30-minute session with a coach to have their baseline lifestyle tracking results explained to them and receive personalised suggestions on lifestyle modifications.
- Experimental group (Experimental): The activities during health screening before the study and at the end of study is similar to the control. Individuals are provided with an educational brochure upon receiving their screening results. Participants will then go through a baseline lifestyle tracking session using a study-issued smartphone and smartwatch, pre-installed with certain study applications, which will be used for the lifestyle tracking sessions. The experimental arm will go through 4 additional lifestyle tracking sessions (i.e., total of 5 including baseline), of which 1 will include Continuous Glucose Monitoring (CGM) tracking. For this CGM tracking session, participants will receive real-time feedback through the study applications, which will display the CGM trace. The data collected during the lifestyle tracking sessions will be discussed with the participants during 3 face-to-face coaching and 2 tele-coaching sessions, where the participants will develop and implement lifestyle change action plans.
  Interventions: Device: CGM lifestyle tracking and coaching

INTERVENTIONS:
Device: CGM lifestyle tracking and coaching — Participants in the experimental group will go through a total of 5 lifestyle tracking sessions (including baseline), of which 1 will include CGM tracking. For this CGM lifestyle tracking session, experimental group participants will receive real-time feedback through the study applications, which will display the CGM trace.
  The data collected during the lifestyle tracking sessions will be discussed with the participants during 3 face-to-face coaching and 2 tele-coaching sessions, where the participants will develop and implement lifestyle change action plans.
  Arms: Experimental group

SUMMARY:
This study seeks to address two questions. Firstly, how might a suite of interventions and data feedback (activity, diet, mood*, continuous blood glucose) through coaching be effective in influencing behaviour change for individuals at-risk of developing type 2 diabetes? Secondly, what elements of coaching might be extracted for automated implementation in a scalable coach-light model?

DETAILED DESCRIPTION:
Face-to-face health coaching is a common lifestyle intervention for healthy individuals who are at risk of chronic diseases such as diabetes. However, it is highly resource-intensive and has limitations in scaling up to reach wider populations. Advances in technology present opportunities to scale health coaching to the wider population through automation, enabling the delivery of personalised messages for individuals via mobile applications.

In addition, continuous glucose monitoring (CGM) devices could also potentially augment the effectiveness of health coaching by providing coaches with a tool for coachees' self-discovery of their individual physiological responses to lifestyles and modifications such as diet and exercise.

As such, the present study seeks to leverage smart wearable devices (e.g., Bluetooth smartwatches) and CGM devices accompanying a customized mobile application to deliver lifestyle coaching interventions. This suite of lifestyle interventions, including feedback about their own blood glucose levels, aims to influence participant's lifestyles and behaviours through guided self-discovery and face-to-face coaching. This intervention will be compared with a control group to examine its effects on lifestyle change, anthropometric measures and biometric measures. In addition, the findings from this study will contribute to the development of a novel coach-light intervention that can be implemented at a wider population level via Singapore's Health Promotion Board's (HPB) existing programmes and channels.

ELIGIBILITY:
Inclusion Criteria:

1. Singaporean Citizens and Permanent Residents
2. Aged 21 to 55
3. Must be literate in English (i.e. able to read and communicate in English) because the primary mode of communication is English
4. Willing and able to use a smartphone
5. Must be at risk of developing Type 2 Diabetes, defined as:

i) Glycated haemoglobin (HbA1c) - At least 5.7% to 6.5% OR Fasting blood glucose of 6.1 to 6.9mmol/L, AND ii) BMI of at least 20kg/m2

Exclusion Criteria:

1. Non-Singaporean Citizens and Permanent Residents
2. Under age 21 or above age 55
3. Ever diagnosed as Type 1 or Type 2 Diabetic (does not include previously diagnosed GDM)
4. Pregnant or planning to be pregnant in the next 6 months or lactating
5. History of skin allergies
6. Taking medications that are known to alter blood sugar levels/ glucose tolerance e.g.

glucocorticoids g) History of mental illness/conditions h) Work requirement that does not allow the carrying of electronic devices (e.g., phone and smartwatch) i) Frequent overseas travelling (e.g., more frequently than once a month, daily or weekly commuting across borders etc.)

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Behaviour, self-efficacy and attitudes | Baseline and at month 3
  Change in behaviour, self-efficacy and attitudes towards diet and exercise from baseline to 3rd month

SECONDARY OUTCOMES:
HbA1c concentration | Baseline and at month 3
  Change in fasting plasma HbA1c concentration from baseline to 3rd month
Plasma glucose concentration | Baseline and at month 3
  Change in fasting plasma glucose concentration from baseline to 3rd month
BMI | Baseline and at month 3
  Change in BMI from baseline to 3rd month
Lipid profile | Baseline and at month 3
  Change in lipid profile from baseline to 3rd month
Systolic and Diastolic Blood pressure | Baseline and at month 3
  Change in systolic and diastolic blood pressure from baseline to 3rd month

CONTACTS AND LOCATIONS:
Overall Officials: Falk Müller-Riemenschneider, Principal Investigator — National University of Singapore
Locations (1):
- Saw Swee Hock School of Public Health, National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dunkley AJ, Bodicoat DH, Greaves CJ, Russell C, Yates T, Davies MJ, Khunti K. Diabetes prevention in the real world: effectiveness of pragmatic lifestyle interventions for the prevention of type 2 diabetes and of the impact of adherence to guideline recommendations: a systematic review and meta-analysis. Diabetes Care. 2014 Apr;37(4):922-33. doi: 10.2337/dc13-2195. PMID 24652723
- [Background] Fukuoka Y, Gay CL, Joiner KL, Vittinghoff E. A Novel Diabetes Prevention Intervention Using a Mobile App: A Randomized Controlled Trial With Overweight Adults at Risk. Am J Prev Med. 2015 Aug;49(2):223-37. doi: 10.1016/j.amepre.2015.01.003. Epub 2015 May 30. PMID 26033349
- [Background] Block G, Azar KM, Romanelli RJ, Block TJ, Hopkins D, Carpenter HA, Dolginsky MS, Hudes ML, Palaniappan LP, Block CH. Diabetes Prevention and Weight Loss with a Fully Automated Behavioral Intervention by Email, Web, and Mobile Phone: A Randomized Controlled Trial Among Persons with Prediabetes. J Med Internet Res. 2015 Oct 23;17(10):e240. doi: 10.2196/jmir.4897. PMID 26499966
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527